CLINICAL TRIAL: NCT03928496
Title: Abobotulinumtoxina Efficacy in Post-Traumatic Headache
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Zirovich0002
Record Dates: First submitted 2019-04-18; First posted 2019-04-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Post-Traumatic Headache
MeSH Terms: conditions — Post-Traumatic Headache | interventions — abobotulinumtoxinA; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The project statistician used a computer-based random number generator to create a randomized treatment allocation schedule that was provided to the pharmacist and nurse practitioner who did not disclose this information. The pharmacist provided the nurse practitioner with the medication in an unlabeled bag, which either included BoNT-A or Normal Saline. Patients were randomized to receive BoNT-A or Normal Saline as first injection. The nurse practitioner reconstituted the medication in a separate room and then provided the investigator with unlabeled syringes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Abobotulinumtoxina (Experimental): 300 units of abobotulinumtoxinA was reconstituted with 2.4 ml of 0.9% preservative free sterile saline so that each 0.1 ml contained 12.5 units of Abobotulinumtoxina 0.1 ml were injected into 31 sites of the head and neck
  Interventions: Drug: AbobotulinumtoxinA
- Placebo (Placebo Comparator): 0.9% preservative free sterile saline. 0.1 ml were injected into 31 sites of the head and neck
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: AbobotulinumtoxinA — Subjects were injected with 0.1 ml (12.5 units of Abobotulinumtoxina) into 31 distinct muscle locations in the head and neck
  Other Names: Dysport
  Arms: Abobotulinumtoxina
Drug: Normal saline — Subjects were injected with 0.1 ml of preservative free normal saline into 31 distinct muscle locations in the head and neck
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy of abobotulinumtoxina on Veterans with post-traumatic headache

DETAILED DESCRIPTION:
A significant proportion of headaches occur following head trauma, and therefore are referred to as post-traumatic headaches (PTH). Traumatic brain injury (TBI) is highly prevalent in the Operation Iraqi Freedom/Operation Enduring Freedom (OIF/OEF) population and consequently there has been a rise in PTH in the clinical setting at VA hospitals. Botulinum toxin type A (BoNT-A) has been shown to be effective in treating chronic migraine and chronic daily headache. It is therefore reasonable to predict that BoNT-A may also be effective in treating PTH. This study proposes that PTH and its associated symptoms may respond positively to BoNT-A treatment due to its similar pathophysiology and clinical resemblance to other headache disorders including tension type headache, typical migraine with or without aura, and chronic daily headache.

Study Design: Veterans with mild, moderate or severe brain injury with a headache developing within 7 days after head trauma and persisting greater than 3 months were recruited from the Veterans Affairs Greater Los Angeles Healthcare System. The study is a prospective, double-blind, randomized, placebo-controlled, cross-over trial.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* age 18-65
* meets International Classification Headache Disorders II (ICHD-II) criteria for post-traumatic headache
* average pain score of greater than 4/10 in severity on the numerical rating system
* Rancho Los Amigos cognitive scale score greater than seven.

Exclusion Criteria:

* Uncontrolled medical condition other than PTH
* Severe additional chronic pain complaint which could not be distinguished from headache pain
* pregnancy, breast feeding,
* prior treatment with botulinum toxin within one year of enrollment
* current substance abuse/dependence
* medical condition that would increase risk of neuromuscular junction blockade with botulinum toxin (myasthenia gravis, Eaton Lambert, amyotrophic lateral sclerosis)
* poorly controlled psychiatric
* initiation of a new anti-depressant or anti-seizure medication within three months of enrolling in study
* ongoing disability or litigation claim.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2017-02-02 (Actual); Study Completion 2017-02-02 (Actual)

PRIMARY OUTCOMES:
Incidence of headaches from baseline | evaluation from time of injection until completion of 12 week follow-up
  Evaluation in weekly incidence of headaches from baseline based on headache diary or weekly phone follow-up

SECONDARY OUTCOMES:
Intensity of headache pain | evaluation from time of injection until completion of 12 week follow-up
  Evaluation of pain intensity using score of headache on Numerical Rating Scale (NRS) over time. The NRS is an 11-point scale for patient self-reporting of pain with 0 being no pain and 10 being the most severe pain.
Number of headache days per week | evaluation from time of injection until completion of 12 week follow-up
  Evaluation of the number of days a headache was present over each week

CONTACTS AND LOCATIONS:
Overall Officials: Milena Zirovich, MD, Principal Investigator — VA Greater Los Angeles
Locations (1):
- VA Greater Los Angeles Healthcare System, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified dataset may be provided upon request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting at 3 months following publication and up to 3 years after publication
Access Criteria: Data access requests will be reviewed and requestors will sign a data access agreement